CLINICAL TRIAL: NCT05818137
Title: A Phase 3 Non-randomized, Non-controlled, Open Label Clinical Study to Evaluate the Efficacy and Safety of MK-7962 (Sotatercept) add-on to Background Therapy in Japanese Participants With Pulmonary Arterial Hypertension (PAH)
Brief Title: A Study of Sotatercept in Japanese Pulmonary Arterial Hypertension (PAH) Participants (MK-7962-020)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7962-020; jRCT2031230046 (Registry Identifier: jRCT); MK-7962-020 (Other: MSD)
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ACE-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sotatercept (Experimental): Participants on background PAH therapy will receive sotatercept subcutaneous (SC) injections at a starting dose of 0.3 mg/kg with a target dose of 0.7 mg/kg every 3 weeks up to 24 weeks. Thereafter, participants may choose to receive the sotatercept treatment at same dose and schedule in the extension treatment period from Week 24 until up to 6 months after sotatercept becomes locally commercially available and reimbursed in Japan.
  Interventions: Biological: Sotatercept

INTERVENTIONS:
Biological: Sotatercept — SC injection at a starting dose of 0.3 mg/kg with a target dose of 0.7 mg/kg every 21 days plus background PAH therapy.
  Other Names: MK-7962; ActRIIA-IgG1Fc; ACE-011

SUMMARY:
This local Phase 3 study is planned to confirm the efficacy and safety in Japanese PAH participants. The primary population of this study is Japanese PAH participants with World Health Organization Functional Class (WHO FC) II or III while the study includes PAH participants with WHO FC I or IV as other populations. There are no hypotheses for this study.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnostic right heart catheterization (RHC) at any time prior to screening confirming the diagnosis of World Health Organization (WHO) pulmonary arterial hypertension (PAH) Group 1 in any of the following subtypes:

  * Idiopathic PAH
  * Heritable PAH
  * Drug/toxin-induced PAH
  * PAH associated with connective tissue disease
  * PAH associated with simple, congenital systemic-to-pulmonary shunts at least 1 year following repair
* PAH classified as WHO functional class (FC) I or symptomatic PAH classified as WHO FC II to IV
* On stable doses of background PAH therapy and diuretics (if applicable) for at least 90 days prior to screening

Exclusion Criteria

* Diagnosis of PH WHO Groups 2, 3, 4, or 5
* Diagnosis of the following PAH Group 1 subtypes:

  * Human immunodeficiency virus (HIV)-associated PAH
  * PAH associated with portal hypertension
  * Schistosomiasis-associated PAH
  * PAH with features of significant venous/capillary pulmonary veno-occlusive disease/pulmonary capillary hemangiomatosis (PVOD/PCH) involvement
* Is on the waiting list for lung transplant
* Pregnant or breastfeeding women
* History of full or partial pneumonectomy
* Pulmonary function test (PFT) values of forced vital capacity (FVC) < 60% predicted at the screening visit or within 6 months prior to the screening visit.
* Initiation of an exercise program for cardiopulmonary rehabilitation within 90 days prior to the screening visit or planned initiation during the study.
* History of more than mild obstructive sleep apnea that is untreated
* Known history of portal hypertension or chronic liver disease, including hepatitis B and/or hepatitis C (with evidence of recent infection and/or active virus replication), defined as mild to severe hepatic impairment.
* History of restrictive, constrictive, or congestive cardiomyopathy.
* History of atrial septostomy within 180 days prior to the screening visit.
* Personal or family history of long QT syndrome (LQTS) or sudden cardiac death.
* Left ventricular ejection fraction (LVEF) < 45% on historical Echocardiogram (ECHO) within 6 months prior to the screening visit.
* Any symptomatic coronary disease events within 6 months prior to the screening visit.
* Cerebrovascular accident within 3 months prior to the screening visit.
* Significant (≥ 2+ regurgitation) mitral regurgitation or aortic regurgitation valvular disease, mitral stenosis and more than mild aortic valve stenosis.
* Prior exposure to sotatercept or luspatercept or history of allergic or anaphylactic reaction or hypersensitivity to recombinant proteins or excipients in investigational product
* Received intravenous inotropes (e.g., dobutamine, dopamine, norepinephrine, vasopressin) within 30 days prior to the screening visit
* Currently enrolled in or have completed any other investigational product study within 30 days
* Weight at the screening is over 85 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2025-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (17):
- Japan (17):
  - Nagoya University Hospital ( Site 2010), Nagoya, Aichi-ken
  - Chiba Saiseikai Narashino hospital ( Site 2004), Narashino, Chiba
  - Kurume University Hospital ( Site 2014), Kurume, Fukuoka
  - Kure Kyosai Hospital ( Site 2017), Kure, Hiroshima
  - Sapporo Medical University Hospital ( Site 2018), Sapporo, Hokkaido
  - Hokkaido University Hospital ( Site 2001), Sapporo, Hokkaido
  - Kobe University Hospital ( Site 2012), Kobe, Hyōgo
  - Tohoku University Hospital ( Site 2002), Sendai, Miyagi
  - National Cerebral and Cardiovascular Center ( Site 2011), Suita, Osaka
  - Hamamatsu University Hospital ( Site 2016), Hamamatsu, Shizuoka
  - The University of Tokyo Hospital ( Site 2006), Bunkyo-ku, Tokyo
  - Kyorin University Hospital ( Site 2005), Mitaka, Tokyo
  - Chiba University Hospital ( Site 2003), Chiba
  - Kyushu University Hospital ( Site 2015), Fukuoka
  - National Hospital Organization Okayama Medical Center ( Site 2013), Okayama
  - International University of Health and Welfare Mita Hospital ( Site 2008), Tokyo
  - Keio university hospital ( Site 2007), Tokyo

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All allocated participants.
Groups:
- Sotatercept: Participants on background PAH therapy received sotatercept subcutaneous (SC) injections at a starting dose of 0.3 mg/kg with a target dose of 0.7 mg/kg every 3 weeks up to 24 weeks. Thereafter, participants received sotatercept at the same dose and schedule in the extension treatment period Week 24 to Week 42.
Period: Primary Treatment Period
Arm/Group | Sotatercept
Started | 46
Completed | 46
Not Completed | 0
Period: Extension Treatment Period
Arm/Group | Sotatercept
Started | 45 (One participant discontinued the study after completing the primary treatment period at Week 24. This participant did not start the extension treatment period.)
Completed | 0
Not Completed | 45
Not completed — Withdrawal by Subject | 1
Not completed — Ongoing participants | 44

BASELINE CHARACTERISTICS:
Population: All allocated participants.
Arm/Group | Sotatercept
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.7 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 46
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Pulmonary Vascular Resistance (PVR) at Baseline [Count of Participants; unit: Participants] — PVR was the resistance against blood flow from the pulmonary artery to the left atrium. PVR was measured by right heart catheterization (RHC). PVR was categorized as ≤800 dyn*sec/cm^5 and >800 dyn*sec/cm^5.
  Participants
    ≤800 dyn*sec/cm^5 | 43
    >800 dyn*sec/cm^5 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Pulmonary Vascular Resistance (PVR) From Baseline at Week 24
Description: PVR was the resistance against blood flow from the pulmonary artery to the left atrium. PVR was measured in dyn*sec/cm^5 by right heart catheterization (RHC). RHC was performed during the screening period (baseline) and Week 24. Per protocol, the change in PVR from baseline at Week 24 was reported for the primary treatment period.
Time Frame: Baseline and Week 24
Population: All participants who received at least one dose of study intervention in the primary treatment period.
Measure: Median (Full Range); unit: dynes*sec/cm^5
Groups:
- Sotatercept - Primary Treatment Period: Participants on background PAH therapy received sotatercept subcutaneous (SC) injections at a starting dose of 0.3 mg/kg with a target dose of 0.7 mg/kg every 3 weeks up to 24 weeks.
Arm/Group | Sotatercept - Primary Treatment Period
Number analyzed (Participants) | 46
dynes*sec/cm^5 | 417.2 [235.2 to 812.8]
Statistical Analysis 1: Comparison: Sotatercept - Primary Treatment Period; Test type: Other; Change from baseline estimate = -99.2, 95% CI 2-sided [-129.6 to -68.4] — The change from baseline estimate and associated 95% confidence interval (CI) based on the Hodges-Lehmann method

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Per protocol, the number of participants who experienced an AE were reported for the primary treatment period.
Time Frame: Up to ~24 weeks
Population: All participants who received at least one dose of study intervention in the primary treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept - Primary Treatment Period
Number analyzed (Participants) | 46
Participants | 43

3. Primary Outcome: Number of Participants Who Discontinued Study Intervention Due to AEs
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Per protocol, the number of participants who discontinued study treatment due to AEs were reported for the primary treatment period.
Time Frame: Up to ~24 weeks
Population: All participants who received at least one dose of study intervention in the primary treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept - Primary Treatment Period
Number analyzed (Participants) | 46
Participants | 0

4. Secondary Outcome: Change From Baseline in Six-Minute Walk Distance (6MWD) at Week 24
Description: The 6MWD was the distance walked in 6 minutes as a measure of functional capacity was measured during the screening period (baseline) and at Week 24. This was assessed using the 6-minute walk test (6MWT). Per protocol, the change from baseline in 6MWD at Week 24 was reported for the primary treatment period.
Time Frame: Baseline and Week 24
Population: All participants who received at least one dose of study intervention in the primary treatment period.
Measure: Median (Full Range); unit: Meter
Arm/Group | Sotatercept - Primary Treatment Period
Number analyzed (Participants) | 46
Meter | 462.0 [305.0 to 560.0]
Statistical Analysis 1: Comparison: Sotatercept - Primary Treatment Period; Test type: Other; Change from baseline estimate = 41.8, 95% CI 2-sided [27.8 to 55.5] — The change from baseline estimate and associated 95% confidence interval (CI) based on the Hodges-Lehmann method

5. Secondary Outcome: Percentage of Participants With Improvement in World Health Organization Functional Class (WHO FC) at Week 24
Description: The severity of participant's pulmonary arterial hypertension (PAH) symptoms will be graded using the WHO FC system. WHO functional classification for PAH ranges from Class I (no limitation in physical activity, no dyspnea with normal activity), Class II (slight limitation of physical activity), Class III (marked limitation of physical activity) and Class IV (cannot perform a physical activity without any symptoms, dyspnea at rest). Participants who improve in WHO FC were classified into "Improved", "No change" and "Worsened". Improvement = reduction in FC, worsened = increase in FC and no change = no change in FC. Per protocol, the percentage of participants with improvement in WHO FC at Week 24 were presented for the primary treatment period.
Time Frame: Baseline and Week 24
Population: All participants who received at least one dose of study intervention in the primary treatment period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sotatercept - Primary Treatment Period
Number analyzed (Participants) | 46
Percentage of participants | 19.6 [9.4 to 33.9]

6. Secondary Outcome: Change From Baseline in N-terminal proB-type Natriuretic Peptide (NT-proBNP) at Week 24
Description: NT-proBNP is an established marker of ventricular dysfunction in participants with PAH. NT-proBNP was measured at Day 1 (baseline) and at Week 24. The change from baseline in NT-proBNP at Week 24 was reported for the primary treatment period.
Time Frame: Baseline and Week 24
Population: All participants who received at least one dose of study intervention in primary treatment period.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Sotatercept - Primary Treatment Period
Number analyzed (Participants) | 46
pg/mL | 18.5 [18.5 to 1471.0]
Statistical Analysis 1: Comparison: Sotatercept - Primary Treatment Period; Test type: Other; Change from baseline estimate = -48.5, 95% CI 2-sided [-77.0 to -24.8] — The change from baseline estimate and associated 95% confidence interval (CI) based on the Hodges-Lehmann method

ADVERSE EVENTS:
Time Frame: Up to approximately 42 weeks (Primary treatment period: Weeks 1-24 & extension Treatment Period: Weeks 24-42)
Description: All-cause mortality was reported on all allocated participants. Serious and nonserious AEs were reported in all participants who received a dose of study intervention.
Groups:
- Sotatercept - Extension Treatment Period: Participants on background PAH therapy received sotatercept subcutaneous (SC) injections at a starting dose of 0.3 mg/kg with a target dose of 0.7 mg/kg every 3 weeks from Week 24 to Week 42.
Arm/Group | Sotatercept - Primary Treatment Period | Sotatercept - Extension Treatment Period
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45
Serious Adverse Events (participants affected / at risk) | 6/46 | 2/45
Other Adverse Events (participants affected / at risk) | 36/46 | 12/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept - Primary Treatment Period (N=46) | Sotatercept - Extension Treatment Period (N=45)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Device physical property issue (Product Issues) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept - Primary Treatment Period (N=46) | Sotatercept - Extension Treatment Period (N=45)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Malaise (General disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 14 (15) | 7 (8)
Haemoglobin increased (Investigations) | 8 (8) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 10 (10) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT05818137/Prot_SAP_000.pdf